CLINICAL TRIAL: NCT03508128
Title: Evaluation of Surgical Electromagnetic Interference in Medtronic Micra Leadless Pacemaker
Brief Title: Evaluation of EMI in Patients With Micra Leadless Pacemaker
Status: Completed | Type: Observational
Sponsor: Edward-Elmhurst Health System (Other)
Responsible Party: Principal Investigator, Janet Gifford, Nurse Practitioner, Edward-Elmhurst Health System
Other Study IDs: EdwardH
Record Dates: First submitted 2018-04-05; First posted 2018-04-25 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Electromagnetic Interference
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Micra subjects: Surgical procedure
  Interventions: Other: surgical procedure

INTERVENTIONS:
Other: surgical procedure — Surgical procedure

SUMMARY:
Subjects with Medtronic Micra leadless pacemaker who require surgical procedures will have postoperative interrogations reviewed for evidence of electromagnetic interference (EMI).

DETAILED DESCRIPTION:
Patients with pacemakers have a potential risk of EMI from sources including electrosurgery which can cause oversensing, pacing inhibition and device reset. There is limited data on surgical EMI in Medtronic Micra leadless pacemakers. The goal of this study is to evaluate for surgical EMI in subjects with leadless pacemakers.

Subjects with Micra leadless pacemakers requiring surgery will have procedure records reviewed for type of procedure and use of electrosurgery. Next postoperative device interrogation will be reviewed for evidence of EMI. EMI will be evaluated by review of sensing integrity counter, heart rate histograms and device reset.

ELIGIBILITY:
Inclusion criteria:

* subjects with an implanted Micra pacemaker who required a surgical procedure

Exclusion Criteria:

* no Micra pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Micra leadless pacemakers implanted at Edward-Elmhurst Healthcare since May 2016 who then required a surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

PRIMARY OUTCOMES:
EMI | up to 6 months next postop interrogation
  Number of subjects with evidence of EMI determined by sensing integrity counter and heart rate histograms

SECONDARY OUTCOMES:
Device reset | up to 6 months next postop interrogation
  Number of subjects with change in programmed parameters showing device reset VVI 65 5V@.4ms

CONTACTS AND LOCATIONS:
Overall Officials: Janet Gifford, MSN, Principal Investigator — Edward-Elmhurst Health
Locations (1):
- EdwardElmhurst Healthcare, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided